CLINICAL TRIAL: NCT01164982
Title: An Open Non-controlled Proof of Concept Investigation Evaluating the Handling of a Soft Silicone Wound Contact Layer, Mepitel® One Used in Acute Wounds in Home Care
Brief Title: Investigation Evaluating Handling of Mepitel® One Used in Acute Wounds in Home Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No resources available at the clinic
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Jenny Thorell, Molnlycke Health Care AB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MPTO 02
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2010-12

CONDITIONS: Acute Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Mepitel One — Each subject will be followed once a week for 3 weeks or until healing if that occurs earlier

SUMMARY:
The primary objective is to evaluate the handling of Mepitel® One when used in acute wounds in home care.

Secondary objective is to evaluate the comfort, conformability, stay-on ability, pain at removal, transparency of dressing and adverse events.

DETAILED DESCRIPTION:
The investigation is designed as an open, non-controlled, proof of concept investigation. Subjects with acute wounds at one centre will be included. Each subject will be followed once a week for 3 weeks or until healing if that occurs earlier. All dressing changes will be done according to clinical routine and registered in a dressing log. Cover dressing will be used when needed according to clinical routine.

A total of 10 subjects will be enrolled provided that they fulfil all the inclusion criteria and none of the exclusion criteria and have signed and dated the written informed consent.

The subjects will be consecutively allocated to a subject code.

At baseline, subject characteristics will be registered together with subject status of health, wound history and wound status, wound characteristics and current treatment of the wound.

The following variables will be measured as follows:

ELIGIBILITY:
Inclusion Criteria:

1. Acute wounds/burns
2. Male or female, 18 years and above, both in- and outpatients.
3. Signed Informed Consent Form

Exclusion Criteria:

1. Wound size above 21x24.5 cm
2. Subject not expected to follow the investigation procedures
3. Subjects previously included in this investigation
4. Subjects included in other ongoing clinical investigation at present or during the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
to evaluate the handling of Mepitel® One when used in acute wounds in home care. | once a week for 3 weeks or until healing

SECONDARY OUTCOMES:
to evaluate the comfort, conformability, stay-on ability, pain at removal, transparency of dressing and adverse events. | once a week for 3 weeks or until healing

CONTACTS AND LOCATIONS:
Overall Officials: Hans J Höning, Dr, Principal Investigator — Chir-Praxis, Hamburg
Locations (1):
- Chir-Praxis, Hamburg, Hamm, Germany